CLINICAL TRIAL: NCT06963788
Title: Double-blind Interventional Study in Southern Vietnam: the Comparative Effects of Using 0.12% Chlorhexidine and Silver Nanoparticles Mouthwashes in Medical Students
Brief Title: The Comparative Effects of Using 0.12% Chlorhexidine and Silver Nanoparticles Mouthwashes in Medical Students
Acronym: mouthwash
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23.134.SV/PCTHĐĐĐ; 23.KR.005 (Other: Can Tho University of Medicine and Pharmacy)
Record Dates: First submitted 2025-04-15; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Dental Plaque and Gingivitis
Keywords: preventative dentistry; dental plaque; mouthwash
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Control group) (Placebo Comparator): This group uses 0.9% sodium chloride
  Interventions: Drug: 0,9% Chloride Sodium
- Group II (Active Comparator): This group uses 0.12% CHX mouthwash
  Interventions: Drug: Chlorhexidine 0,12%
- Group III (Active Comparator): This group uses AgNPs mouthwash
  Interventions: Drug: Silver nanoparticles mouthwash

INTERVENTIONS:
Drug: Chlorhexidine 0,12% — Rinse mouth with 10ml for 30 seconds after brushing teeth for 30 minutes
  Other Names: CHX mouthwash
  Arms: Group II
Drug: 0,9% Chloride Sodium — Rinse mouth with 10ml for 30 seconds after brushing teeth for 30 minutes
  Other Names: NaCl 0,9%
  Arms: Group I (Control group)
Drug: Silver nanoparticles mouthwash — Rinse mouth with 10ml for 30 seconds after brushing teeth for 30 minutes
  Other Names: AgNPs mouthwash
  Arms: Group III

SUMMARY:
This double-blind, randomized intervention study aims to evaluate and compare the efficacy of 0.12% Chlorhexidine (CHX) mouthwash and Nano Silver (AgNPs) mouthwash. Specifically, it seeks to address the following research questions:

How effective are 0.12% CHX and AgNPs mouthwashes in controlling dental plaque accumulation, reducing gingival inflammation, and maintaining salivary pH balance?

How do these two mouthwashes compare in terms of relevant clinical parameters?

The study design includes three groups: Group I (control), which will receive 0.9% sodium chloride (saline solution); Group II, which will receive 0.12% CHX mouthwash; and Group III, which will receive AgNPs mouthwash. Participants will be selected based on defined inclusion and exclusion criteria.

Subjects will be randomly assigned to one of the three groups, ensuring an even distribution of male and female participants. Clinical parameters will be recorded at baseline and after 21 days of intervention. These parameters include the Gingival Index (GI), the Quigley-Hein Plaque Index (QHI), microbial colony counts, and salivary pH levels.

Blinding was maintained throughout the study: neither participants nor clinical evaluators were aware of group assignments. The individual responsible for coding the mouthwash formulations was not involved in any other part of the study and disclosed the codes only after data analysis was completed.

DETAILED DESCRIPTION:
Sample collection procedure Before the study, participants underwent a comprehensive oral health screening to evaluate dental caries, inflammation, and other dental conditions. Participants were instructed to fast for 2 hours prior to the examination to ensure accurate results. The selection was based on specific inclusion and exclusion criteria, and baseline clinical characteristics were accurately recorded. At baseline (day 0), a detailed assessment of microbial counts was conducted. Saliva samples were cultured on agar plates with standardized volumes of 10 µL, diluted to concentrations of 1/100 and 1/1000. After incubation at 37°C for 24 hours, colony-forming units (CFUs) were counted, and the microbial density was calculated per milliliter of saliva, then converted to a logarithm (CFU/mL) for statistical analysis. Additionally, saliva pH was measured using a calibrated digital pH meter, equipped with an electrode and a temperature sensor (Hanna HI2211-02 Benchtop pH Meter, Italy). The level of plaque was assessed using the QHI. After 21 days of use (day 21), a reassessment was conducted to reflect the processes from day 0, including the reevaluation clinical parameters such as GI, QHI, microbial counts, and saliva pH Statistical analysis The assembled data were imported into Microsoft Excel 2020 and Google Drive software, followed by SPSS Statistics 22.0 for analysis and accomplishment he ANOVA, paired T-tests, and Tukey post-hoc tests were employed to analyze the study parameters at baseline and after 21 days of using mouthwash.

Study error The total number of colonies formed was counted and analyzed by a microbiologist. For parameters such as GI, QHI, and salivary pH, assessments were performed by a dentist. Investigators were blinded to the group assignments of the samples. The microbiologist's consistency was evaluated as follows: after the initial sample measurements were taken, 30 randomly selected samples were re-evaluated using the same method by the same individual (reproducibility test), approximately 30 minutes later. Similarly, the consistency of the dentist was assessed. Data from the second measurement were compared with the first using Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible for inclusion if they met all of the following conditions:

* Had not used systemic antibiotics, corticosteroids, or mouthwash for at least 28 days prior to the start of the study;
* Maintained stable oral and general health throughout the study period.

Exclusion Criteria:

Participants were excluded from the study if they met any of the following conditions:

* Had incomplete data or demonstrated non-compliance with study protocols;
* Presented with active oral infections;
* Were undergoing ongoing orthodontic or cosmetic dental treatments;
* Had systemic conditions such as autoimmune disorders, diabetes mellitus, hypertension, hematological diseases, or psychiatric disorders.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Plaque Control Effectiveness After 21 Days of Use Between Two Types of Mouthwash: Chlorhexidine 0.12% and Silver Nanoparticles | From the initiation of mouthwash use on Day 1 until the completion of the intervention on Day 21
  Measurement Tool: Quigley-Hein Plaque Index (QHI)
  Measurement Tool Description:
  The Quigley-Hein Plaque Index (QHI) is a smooth surface index that assesses dental plaque by staining the plaque with a disclosing agent and categorizing it into six grades based on severity:
  Grade 0: No plaque present.
  Grade 1: Isolated islands of plaque.
  Grade 2: A clearly defined continuous plaque line at the gingival margin, extending up to 1 mm.
  Grade 3: Plaque covering the cervical third of the tooth.
  Grade 4: Plaque covering up to the middle third of the tooth.
  Grade 5: Plaque extending beyond the middle third and reaching the incisal or occlusal edge.
  Index Calculation:
  QHI is calculated by summing the severity grades and dividing by the total number of teeth evaluated, as follows:
  QHI = the severity levels/ Number of teeth used for evaluation
Comparison of the Effectiveness of Reducing Gingivitis After 21 Days of Use Between Two Mouthwashes: Chlorhexidine 0.12% and Silver Nanoparticles | From the initiation of mouthwash use on Day 1 until the completion of the intervention on Day 21
  Measurement Tool: Gingival Index (GI)
  Description of the Measurement Tool:
  The presence of gingivitis was assessed using a periodontal probe and evaluated according to the Gingival Index (GI). The severity of gingival inflammation was categorized into four grades:
  Grade 0: Normal gingiva, with no signs of inflammation.
  Grade 1: Mild gingivitis, characterized by slight color changes and mild swelling of the gingiva, without bleeding upon probing.
  Grade 2: Moderate gingivitis, with redness, swelling, a shiny surface appearance, and bleeding upon gentle probing.
  Grade 3: Severe gingivitis, presenting with marked redness, swelling, ulceration, and spontaneous bleeding.
  The GI score for an individual tooth is determined by averaging the scores from four designated sites (buccal, lingual, mesial, and distal surfaces).
  The overall GI for an individual is calculated as the mean GI score across all examined teeth.
Comparison of the effectiveness of reducing the number of bacteria in saliva after 21 days of use between two mouthwashes: Chlorhexidine 0.12% and silver nanoparticles. | From the initiation of mouthwash use on Day 1 until the completion of the intervention on Day 21
  Method: The number of colonies growing on culture media was determined by counting colony-forming units (CFU).
  Unit of measurement: CFU/mL
Comparison of the effectiveness of pH control in saliva after 21 days of use between two mouthwashes: Chlorhexidine 0.12% and silver nanoparticles | From the initiation of mouthwash use on Day 1 until the completion of the intervention on Day 21
  Saliva pH was measured using a calibrated digital pH meter, equipped with an electrode and a temperature sensor (Hanna HI2211-02 Benchtop pH Meter, Italy)

CONTACTS AND LOCATIONS:
Overall Officials: Thao Do, Assoc. Prof., Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

REFERENCES:
- [Background] Maher Y.A., Fathi A., Sembawa B.A., Elkhyat S.H., Hafiz H.F., et al. Effectiveness of Mouthwash-Containing Silver Nanoparticles on Cariogenic Microorganisms, Plaque Index, and Salivary pH in A Group of Saudi Children. The Open Dentistry Journal, (2022), 16, https://doi.org/10.2174/18742106-v16-e2209090
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684